CLINICAL TRIAL: NCT03956264
Title: Interest of Virtual Reality in the Management of Anxiety and Pain Related to Post-cardiac Surgery Care
Acronym: ARVACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMC Ambroise Paré (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019/01
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2020-08

CONDITIONS: Surgery, Cardiac
Keywords: Pain; Anxiety; Mediastinal drain removal
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — kalinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR (Experimental): VR Installation 5 min before the drain removal and stop 10 min after the procedure.
  If Pain assessed by numerical rating scale (NRS) > 4, administration of morphine.
  Interventions: Device: Virtual Reality
- Kalinox® (Active Comparator): Start of Kalinox® administration by inhalation with a facial mask 1 min before the drain removal and stop after the procedure according to the usual procedure of the service.
  If Pain NRS > 4, administration of morphine.
  Interventions: Drug: Kalinox

INTERVENTIONS:
Device: Virtual Reality — Deepsen offers a VR platform that provides patients with immersive contents aimed to distract, inform, soften and improve the healthcare experience
  Arms: VR
Drug: Kalinox — Gas mixture composed of 50% Nitrous Oxide and 50% Oxygen
  Arms: Kalinox®

SUMMARY:
This study compares Virtual Reality versus Nitrous oxide administration for the management of anxiety and pain related to post-cardiac surgery care, especially during removal of mediastinal drainage.

DETAILED DESCRIPTION:
After cardiac surgery, the mediastinal and pleural drains are usually removed the second postoperative day, in the absence of complications. This procedure, realized by nurses, is a source of anxiety and pain for patients.

Nitrous oxide (Kalinox®) is commonly used to manage many situations of anxiety, including the removal of mediastinal and/or pleural drains, and has shown a greater effect than placebo in this indication.

Virtual Reality (VR) is a recent technology that allows the representation of a pleasant environment in three dimensions with a complete immersion by a helmet. By distracting patients, this technology can reduce anxiety, discomfort and ultimately pain associated with care.

This randomized monocentric trial compares VR versus Kalinox® administration for the management of anxiety and pain related to post-cardiac surgery care, especially mediastinal and/or pleural drain removal.

ELIGIBILITY:
Inclusion Criteria:

* Extubated after cardiac surgery
* Sinus rhythm
* Consent for participation
* Affiliation to the social security system

Exclusion Criteria:

* Pacemaker
* Visual acuity making impossible the use of virtual reality
* Intolerance to morphine
* Contraindication to Kalinox®
* Pregnant or breastfeeding women
* Patients under protection of the adults (guardianship, curators or safeguard of justice)
* Communication difficulties or neuropsychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Assessment of patient comfort | 30 minutes
  Variation of the Analgesia / Nociception Index (ANI)

SECONDARY OUTCOMES:
Level of pain during drain removal | 30 minutes
  Pain numerical rating scale (NRS) ranging from 0 to 10 (0=no pain, 10=worst possible pain)
Level of anxiety during drain removal | 30 minutes
  Anxiety NRS ranging from 0 to 10 (0=no stress, 10=worst possible stress)
Morphine consumption | 1 hour
  Cumulated dose of oxynorm (mg)
Side effects due to Virtual Reality | 2 hours
  Onset of vertigo, nausea or vomiting
Patient satisfaction | 2 hours
  Satisfaction verbal rating scale (VRS) ranging from 0 to 4 (0=unsatisfied, 4=very satisfied)
Health staff satisfaction | 30 minutes
  Satisfaction VRS ranging from 0 to 4 (0=unsatisfied, 4=very satisfied)
Side effects due to Kalinox | 2 hours
  Onset of delirium, euphoria or headache
Correlation between ANI and Pain NRS | 30 minutes
Correlation between ANI and Anxiety NRS | 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- CMC Ambroise Paré, Neuilly-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Laghlam D, Naudin C, Coroyer L, Aidan V, Malvy J, Rahoual G, Estagnasie P, Squara P. Virtual reality vs. Kalinox(R) for management of pain in intensive care unit after cardiac surgery: a randomized study. Ann Intensive Care. 2021 May 13;11(1):74. doi: 10.1186/s13613-021-00866-w. PMID 33983498